CLINICAL TRIAL: NCT06740422
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase Ⅲ Clinical Trial on the Efficacy and Safety of Xuanhuang Runtong Tablet in Treating Constipation (Yin-deficiency Type).
Brief Title: Xuanhuang Runtong Tablet in the Treatment of Constipation (Yin-deficiency Type)
Acronym: XHRT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Shengsheng Zhang, Principal Investigator, Beijing Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XHRT-Ⅲ-2024
Record Dates: First submitted 2024-12-10; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xuanhuang Runtong Tablet group (Experimental): Xuanhuang Runtong Tablet, 4 tablets (1.84 g herb per tablet) per dose, three times a day
  Interventions: Drug: Xuanhuang Runtong Tablet
- Placebo group (Placebo Comparator): Xuanhuang Runtong Tablet Simulator, 4 tablets (0 g herb content per bottle) per dose, three times a day
  Interventions: Drug: Xuanhuang Runtong Tablet Simulator

INTERVENTIONS:
Drug: Xuanhuang Runtong Tablet — A synthetic tablet is mainly composed of Radix Rehmanniae, Radix Scrophulariae, Radix Angelicae Sinensis, Semen Persicae, Herba Cistanches, Fructus Cannabis, Semen Cassiae, Fructus Aurantii Immaturus and Aloe.
  Arms: Xuanhuang Runtong Tablet group
Drug: Xuanhuang Runtong Tablet Simulator — Xuanhuang Runtong Tablet Simulator
  Arms: Placebo group

SUMMARY:
This trial is a randomized, double-blind, placebo-controlled parallel-group, multicenter Phase III clinical trial. It is to evaluate the efficacy and safety of Xuanhuang Runtong Tablets in subjects with constipation (Yin-deficiency type) after 4 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to enter the run-in period:

1. Meeting the diagnostic criteria of traditional Chinese medicine (TCM) constipation;
2. Meeting the TCM syndrome differentiation criteria of constipation with yin deficiency syndrome;
3. Both males and females are eligible, aged between 18 and 70 years old (including 18 and 70);
4. Willing to participate in the trial and sign the informed consent form.

At the end of the run-in period, subjects must meet all of the following criteria to enter the treatment period:

1. Meeting the diagnostic criteria of TCM constipation;
2. Meeting the TCM syndrome differentiation criteria of constipation with yin deficiency syndrome;
3. The number of spontaneous bowel movements in the last week of the run-in period is less than 3.

Exclusion Criteria:

Subjects with any of the following items cannot enter the run-in period/treatment period:

1. Subjects with constipation or severe anal diseases causing defecation disorders diagnosed by researchers due to rectal, colonic organic diseases (such as tumors, inflammatory bowel diseases, intestinal adhesions, colon tuberculosis, etc.);
2. Subjects with constipation caused by central nervous system diseases (such as multiple sclerosis, Parkinson's disease, spinal cord injury, etc.) or muscle diseases (such as amyloidosis, dermatomyositis, etc.) known or identified as being caused by drugs;
3. Subjects with colonoscopy results showing intestinal polyps > 0.5 cm or quantity > 3 (subjects with removed intestinal polyps are not excluded, but those with tubular adenoma accompanied by high-grade intraepithelial neoplasia or those who need to re-examine colonoscopy in the near future are excluded);
4. Subjects who have taken drugs for treating constipation within 1 week before screening or within 5 half-lives (calculated according to the longer time);
5. Subjects with severe heart, liver, kidney, brain, blood, metabolic and endocrine system diseases and unstable conditions requiring drug adjustment at any time, and patients with malignant tumors;
6. Subjects who are evaluated by researchers as unable to cooperate with clinical trialists in terms of psychological, mental status or cognitive ability, language expression ability, etc. or have a history of severe mental illness, such as patients with severe depression and severe anxiety.
7. Subjects who have had abdominal surgery within 3 months before screening or plan to have abdominal surgery during the trial period;
8. Subjects with HbA1c > 8.5% at screening;
9. Subjects with ALT or AST ≥ 1.5 times the upper limit of the normal value, or Scr > the upper limit of the normal value;
10. Subjects with known or suspected allergies or severe adverse reactions to the components of Xuanhuang Runtong Tablets or Bisacodyl Enteric-coated Tablets, or with an allergic constitution (such as allergies to two or more drugs or foods);
11. Subjects who have participated in other clinical trials and taken trial drugs within the past 3 months;
12. Subjects with suspected or confirmed history of alcohol or drug abuse;
13. Pregnant or lactating women; or female and male subjects of childbearing potential who are unwilling or unable to take effective contraceptive measures during the trial period;
14. Subjects with other conditions that researchers consider inappropriate to participate in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Complete Spontaneous Bowel Movement (CSBM) response rate after 4 weeks of treatment. | Examination will be performed 4 weeks of treatment.
  CSBM: The number of spontaneous bowel movements with a complete sense of evacuation without taking rescue laxatives or with the assistance of manipulation. (Taking rescue medications within 24 hours before defecation is not counted as CSBM).
  Weekly response: If a patient has at least 3 CSBMs in a week and an increase of at least 1 CSBM compared to the baseline, it is considered a weekly response.
  CSBM response: The patient meets the CSBM weekly response for at least 50% of the weeks during drug treatment (e.g., 3 out of 4 weeks).
  Overall CSBM response rate = Number of CSBM responders / Total number of observed patients × 100%.

SECONDARY OUTCOMES:
Complete Spontaneous Bowel Movement (CSBM) response rate after 2 weeks of treatment. | Examination will be performed 2 weeks of treatment.
  Overall CSBM response rate = Number of CSBM responders / Total number of observed patients × 100%.
The change in the number of bowel movements (BM) at the last week compared to baseline | Evaluation will be performed at baseline and 4 weeks of treatment.
  The patient recorded the number of BMs every day using a diary card.
The change in the number of spontaneous bowel movements (SBM) at the last week compared to baseline . | Evaluation will be performed at baseline and 4 weeks of treatment.
  The patient recorded the number of SBMs every day using a diary card.
The change in the fecal characteristics score (using the Bristol Stool Form Scale) at the last week compared to baseline. | Evaluation will be performed at baseline and 4 weeks of treatment.
  Bristol Stool Form Scale： Type 1 Separate hard lumps, like nuts. Type 2 Sausage-shaped but lumpy. Type 3 Like a sausage or snake but with cracks on its surface. Type 4 Like a sausage or snake, smooth and soft. Type 5 Soft blobs with clear-cut edges. Type 6 Fluffy pieces with ragged edges, a mushy stool.Type 7 Watery, no solid pieces. The 1-7 types correspond to scores of 1-7 respectively.
The change in the degree of difficulty in passing stools score (using the Likert scale) at the last week compared to baseline. | Evaluation will be performed at baseline and 4 weeks of treatment.
  The Patient Assessment of Constipation Symptoms (PAC-SYM) questionnaire uses a Likert scale grading system for rating the severity of constipation symptoms, which is divided into five levels of severity: 0, 1, 2, 3, and 4.
The proportion of subjects with fecal characteristics of type 4 or 5 in the last spontaneous bowel movement (SBM) during the treatment period. | Evaluation will be performed at baseline and 4 weeks of treatment.
  Calculate the proportion of subjects whose fecal consistency of the last spontaneous bowel movement (SBM) during the treatment period is Type 4 or Type 5 among all subjects.
The changes inTraditional Chinese Medicine (TCM) syndrome scores at the last week compared to baseline. | Examination will be performed at baseline and 4 weeks of treatment.
  The TCM syndrome score of constipation consists of 8 questions, and the total scores are ranging from 0 to 24 with higher scores indicating more severe disease.
Efficacy of TCM syndromes | Examination will be performed at baseline and 4 weeks of treatment.
  The efficacy index of TCM syndromes : (pre - treatment score - post - treatment score) / pre - treatment score × 100%. It is divided into four levels: clinical recovery, marked effectiveness, effectiveness, and ineffectiveness.
The disappearance rate of single symptoms of TCM syndromes | Examination will be performed at baseline and 4 weeks of treatment.
  The disappearance rate of single symptoms of TCM syndromes refers to the percentage of the number of cases with a single - symptom score of 0 in each single symptom among the total number of cases (when calculating the denominator, subjects with a single - symptom score of 0 at baseline need to be excluded).
The use of rescue medication. | Examination will be performed 4 weeks of treatment.
  Calculate the total number of rescue medication doses taken during the treatment period.
Changes in the Patient Assessment of Constipation Quality of Life (PAC-QOL) score compared to baseline at 4 weeks of treatment | Examination will be performed at baseline and 4 weeks of treatment.
  Calculate the total PAC-QOL score and the change in scores for the physiological, psychosocial, worries, and satisfaction domains compared to baseline

IPD SHARING:
Plan to Share IPD: No